CLINICAL TRIAL: NCT01257399
Title: Comparative Efficacy and Safety Study in Patients With Ulcerative Colitis in Remission Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Collaborators: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03010302A; 2007L03525 (Other Grant/Funding Number: SFDA_CTA)
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Ulcerative Colitis in Remission
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asacol® (Experimental): Import Mesalazine
  Interventions: Drug: Asacol®
- Mesalazine (Active Comparator): Marketed Mesalazine
  Interventions: Drug: Mesalazine

INTERVENTIONS:
Drug: Asacol® — 400 mg tablets
  Other Names: Import Mesalazine
  Arms: Asacol®
Drug: Mesalazine — 400mg tablets
  Other Names: Marketed Mesalazine
  Arms: Mesalazine

SUMMARY:
To demonstrate that import Mesalazine (ASACOL®) is non-inferior to the reference drug, marketed Mesalazine, regarding the primary endpoint (rate of non-emergence of bloody stool), in patients with Ulcerative Colitis in remission, treated for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis in remission who are defined to show an Ulcerative Colitis-Disease Activity Index (UC-DAI) score of 2 or less and a bloody stool score of 0.

Exclusion Criteria:

* Patients who take adrenal corticosteroid (oral formulation, enemas, suppository, agents for hemorrhoidal disease, injectable solution) within 14 days before start of administration of clinical study drug.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Rate of non-emergence of bloody stool | Week 48

SECONDARY OUTCOMES:
1) Period of non-emergence of bloody stool, 2) Rate of non-recurrence, 3) Period of non-recurrence, 4) Reduction of UC-DAI score | Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Hospital, Shanghai, China

REFERENCES:
- [Derived] Sun J, Yuan Y. Mesalazine Modified-Release Tablet in the Treatment of Ulcerative Colitis in the Remission Phase: A Chinese, Multicenter, Single-Blind, Randomized Controlled Study. Adv Ther. 2016 Mar;33(3):410-22. doi: 10.1007/s12325-016-0304-y. Epub 2016 Feb 23. PMID 26905266